CLINICAL TRIAL: NCT02688205
Title: Correlation Between Cyriax's Functional Examination and Ultrasound Examination in Patients With Shoulder Pain
Status: Completed | Type: Observational
Sponsor: Shin Kong Wu Ho-Su Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 20140107R; SKH-8302-103-DR-37 (Other Grant/Funding Number: Shin Kong Wu Ho-Su Memorial Hospital)
Record Dates: First submitted 2015-05-15; First posted 2016-02-23 (Estimated); Last update posted 2020-12-23 (Actual); Status verified 2016-02

CONDITIONS: Shoulder Pain
Keywords: Cyriax's functional examination; Ultrasound; Correlation; Resisted test
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Shoulder pain group: The participants receive Cyriax's functional examination after history taking, and will be examined by ultrasound in one week.
  Interventions: Other: Cyriax's functional examination; Device: Ultrasound examination
- Without shoulder pain group: The participants receive Cyriax's functional examination after history taking, and will be examined by ultrasound in one week.
  Interventions: Other: Cyriax's functional examination; Device: Ultrasound examination

INTERVENTIONS:
Other: Cyriax's functional examination — included active range of motion, passive range of motion, resisted test and accessory test for shoulder pain evaluation
Device: Ultrasound examination — to evaluate rotator cuff, acromio-clavicular joint, and subdeltoid-subacromial bursa

SUMMARY:
Shoulder problems cause substantial disability in daily living, work, leisure activity, and exercise. The presence of shoulder problem such as rotator cuff pathology reported was highly predictive of impaired health-related quality of life.

Many tests were used for physical examination of the shoulder. The reliability and validity of the tests have been studied before. However, a systemic review concluded that there was conflicting evidence in reliability of each or combined tests. Functional examination of the shoulder by Cyriax is composed of a series of tests to evaluate a shoulder problem. It includes three arm elevation, three tests for glenohumeral joints, and six resisted tests.

As far as the investigators know, correlation of Cyriax functional examination with the ultrasonographic findings has never been reported before. Therefore, the aim of this study is to compare the clinical diagnosis by Cyriax's functional examination with ultrasound findings in patients with shoulder pain.

DETAILED DESCRIPTION:
There are two groups with fifty patients in each group. First group is patients who have unilateral or bilateral shoulder pain from the outpatient clinic of Department of Physical Medicine and Rehabilitation in Shin Kong Wu Ho-Su Memorial Hospital. The other group is control group who has no shoulder problems. Both groups will receive Cyriax's functional examination of the shoulder after history taking, and will be examined by shoulder ultrasound in one week.

ELIGIBILITY:
Inclusion Criteria:

Study group:

1. patients with unilateral or bilateral shoulder pain with unknown causes;
2. age≥ 20 years old.

Control group:

1. patients without unilateral or bilateral shoulder pain;
2. age≥ 20 years old.

Exclusion Criteria:

1) chronic inflammatory joint disease, infections or tumors of the shoulder, previous fracture or surgery of shoulder, and referred pain from cervical origin or visceral organs.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with or without shoulder pain
Sampling Method: Non-Probability Sample
Enrollment: 206 (Actual)
Dates: Start 2014-03; Primary Completion 2015-06 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Cyriax's functional examination for diagnosis | 1 week
  After Cyriax's functional examination for evaluating shoulder pain, a clinical diagnosis is made by the physician
Ultrasound examination for diagnosis | 1 week
  Ultrasound examination is done in one week after Cyriax's functional examination for detailed shoulder pathology evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Lin-Fen Hsieh, M.D., Principal Investigator — Shin Kong Wu Ho-Su Memorial Hospital
Locations (1):
- Shin Kong Wu Ho-Su Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided